CLINICAL TRIAL: NCT07151261
Title: Effects of Daily Intake of Ashwagandha (Withania Somnifera) Root Extract Sustained Release (SR) Capsules 150mg on Disturbed Sleep: a Phase II, Randomized Placebo-controlled Trial With Wearable Device
Brief Title: Ashwagandha for Nighttime Waking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Joshua Goldenberg, Principal Investigator, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ES43025
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Disturbed Sleep
Keywords: Ashwagandha; Disturbed Sleep; Waking After Sleep Onset; Oura ring
MeSH Terms: conditions — Parasomnias | interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained-Release Ashwagandha Supplement (Experimental): Sustained-release, lower-dosage (150mg) Ashwagandha supplement; 1 capsule 1 time per day.
  Interventions: Dietary Supplement: Ashwagandha
- Placebo (Placebo Comparator): Placebo Supplement: Consists of microcrystalline cellulose and is matched for shape, color, and smell. 1 capsule, 1 time per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ashwagandha — Sustained-Release, lower-dosage (150mg) Ashwagandha Supplement, 1 capsule 1 time per day.
  Other Names: Withania Somnifera
  Arms: Sustained-Release Ashwagandha Supplement
Other: Placebo — This placebo does not contain any of the interventional dietary supplement. The placebo consists of microcrystalline cellulose and is matched for shape, color, and smell. 1 capsule, 1 time per day.
  Arms: Placebo

SUMMARY:
The purpose of this research is to evaluate the effect of a sustained-release, lower-dosage (150mg) Ashwagandha supplement to reduce disturbed sleep. 54 participants, after randomization, will take either an Ashwagandha supplement or a placebo daily for 28 days (week 4) and wear an Oura ring. The Oura ring will measure waking after sleep onset (WASO). Questionnaires to evaluate quality of life and sleep will be administered at baseline and week 4.

DETAILED DESCRIPTION:
Each participant will be in the study for about 5 weeks (1 preparation week and 4 weeks for the trial). Questionnaires consist of the Patient-Reported Outcomes Measurement Information System (PROMIS-29). Subjects will be screened for mild sleep disturbance using the PROMIS Sleep Disturbance questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age: Male and non-pregnant female adult participants must be between 18 and 65 years of age.
* Female subjects of childbearing potential must be using a medically acceptable form of birth control, as there are unknown pregnancy risks when starting any new supplement.
* Female subjects of non-childbearing potential must be amenorrheic for at least 1 year or have had a hysterectomy and/or bilateral oophorectomy.
* Sleep Quality: Otherwise, healthy individuals with a raw score of 25-29 (T-score of approximately 55.0-59.9) on the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 8a, indicating at least mild sleep disturbance.
* Sleep Hygiene: Willing to follow basic sleep hygiene protocols (dark/dim lights, quiet location/white noise, regular sleep routine, abstaining from digital activity 1 hour prior to sleep) during the Baseline week and the 28-day trial.
* Wearable Device: Participants must be willing to comply with study procedures, including wearing the Oura Ring nightly (at least 4 nights per week) and completing questionnaires.
* Informed Consent: Participants must be able to provide informed consent and comply with the study procedure.
* Willing to wear the Oura Ring for a total of 35 days (7-day base + 28 days of trial)
* Willing to maintain current dietary patterns, activity level, and stable body weight for the duration of the study, and refrain from any drastic lifestyle changes.
* Willing to refrain from using sleep-promoting supplements or medications during the study, such as melatonin, antihistamines, valerian root, chamomile, magnesium, and cannabinoids (CBD).
* Results of screening procedures/ lab investigations are within normal range or considered not clinically significant by the Principal Investigator.
* Willing to undergo study procedures including safety lab tests and urine pregnancy test (UPT only for women of childbearing potential).

Exclusion Criteria:

* Age: Participants younger than 18 and older than 65 years of age.
* Use of Medications: Current use of sleep-promoting or sleep-disrupting medications or supplements.
* Diagnosed Sleep Disorder: Sleep apnea, narcolepsy, or other for which they are taking medication.
* Other Conditions: Significant medical or psychiatric conditions that could interfere with sleep assessment.
* Irregular Sleep Schedules: Shift workers or those with irregular sleep schedules, as well as anyone with a newborn or having a lifestyle likely to interfere with sleep patterns (eg: jet lag).
* Pregnancy or Lactation: Individuals who are pregnant, lactating, or planning a pregnancy within the next 30 days.
* Post-menopausal female subjects on any Hormone Replacement Therapy
* Allergies: Known allergy or hypersensitivity to any component of the study product.
* Alcohol Intake: History or presence of excessive alcohol use (> 8 drinks per week in women and > 15 drinks per week in men within the past month) or use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.) or addiction to nicotine (current smokers/tobacco users)
* Chronic Illness: Participants with chronic conditions such as liver disease, kidney disease, or severe cardiovascular disease or cancer, colorectal disease and/or other rare disorders that at the discretion of the Principal Investigator (PI) or Clinical Investigator (CI) may impact their safety or confound trial results
* Other Medications: Subjects taking insulin, psychotropics, anxiolytics, sedatives, hypnotics or herbal supplements / Over the counter (OTC) product / multivitamins etc. for sleep or anxiety or any other psychological condition, or any other prescription product which has a known side effect of causing somnolence or sleep problems, within one month prior to the screening visit.
* High-risk medications: The use of any high-risk medications with narrow therapeutic indices metabolized by cytochrome (CYP450) enzymes: Warfarin (CYP2C9), Tacrolimus/Cyclosporine (CYP3A4), Efavirenz (CYP2B6), and Codeine (CYP2D6).
* Drugs requiring activation for efficacy: Clopidogrel (CYP2C19), Codeine (CYP2D6), and Tamoxifen (CYP2D6).
* Participation in Other Trials: Currently participating in another interventional research study or participated in another interventional research study within 90 days of screening
* Any condition that in opinion of the Investigator, does not justify the Subjects' participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Disturbance: Change from Baseline in the Mean Waking After Sleep Onset (WASO) to Week 4 | From Baseline to Week 4 (28 days)
  WASO is measured nightly in hours and minutes via an Oura Ring. The Oura Ring must be worn at least 4 nights per week on average from Baseline (7 days) + 28 days.
  Primary analysis: Change in WASO will be measured as the average of the final 4 days of Week 4 minus the average WASO of the Baseline Week.
  Secondary analysis: Change in WASO will be measured as the average of Week 4 minus the average WASO of the Baseline Week.

SECONDARY OUTCOMES:
Change from Baseline in the Mean Patient-Reported Outcomes Measurement Information System (PROMIS-29) Sleep Disturbance Subdomain to Week 4 | From Baseline to End of Week 4 (28 days)
  Subjective sleep disturbance measured via the PROMIS-29 Profile v2.0 Sleep Disturbance Subdomain. The raw sleep disturbance summed scores range from 4 to 20, with T-scores ranging 32.0 to 73.3, respectively. For Sleep Disturbance, higher scores indicate worse health than average.
  For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
  The sleep quality question is measured as 1 "Very Good" to 5 "Very Poor." The sleep refreshing question is measured as 1 "Very Much" to 5 "Not at all." The two remaining questions problem with sleep and difficulty with sleep are both measured as 1 "Not at all" to 5 "Very Much."
Change from Baseline in Mean PROMIS-29 Sleep Quality Question to Week 4 | From Baseline to End of Week 4 (28 days)
  Sleep quality measured via the PROMIS-29 Sleep Quality question. Scores range from 1 "Very Good" to 5 "Very Poor"

OTHER OUTCOMES:
Change from Baseline in the Mean PROMIS-29 Fatigue Subdomain to Week 4 | Baseline to End of Week 4 (28 days)
  Subjective Fatigue measured via the PROMIS-29 Profile v2.0 Fatigue Subdomain. The raw fatigue summed scores range from 4 to 20, with T-scores ranging 33.7 to 75.8, respectively. For Fatigue, higher scores indicate worse health than average.
  For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
  All four fatigue questions are measured as 1 "Not at all" to 5 "Very much."
Change from Baseline in the Mean PROMIS-29 Anxiety Subdomain to Week 4 | From baseline to End of Week 4 (28 days)
  Subjective anxiety measured via the PROMIS-29 Profile v2.0 Anxiety Subdomain. The anxiety summed scores range from 4 to 20, with T-scores ranging from 40.3 to 81.6, respectively. For Anxiety, higher scores indicated worse health than average.
  For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
  All four anxiety questions are measured as 1 "Never" to 5 "Always."
Change from Baseline in the Mean PROMIS-29 Depression Subdomain to Week 4 | From Baseline to Week 4 (28 days)
  Subjective depression measured via the PROMIS-29 Profile v2.0 Depression Subdomain. The raw depression summed scores range from 4 to 20, with T-scores ranging from 41.0 to 79.4, respectively. For Depression, higher scores indicate worse health than average.
  For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
  All four depression questions are measured as 1 "Never" to 5 "Always."
Change from Baseline in the Mean Sleep Onset Latency (SOL) to Week 4 | From Baseline to Week 4 (28 days)
  SOL is measured objectively via an Oura Ring in seconds. SOL is measured from the local time when the sleep period started, based on the connected mobile device clock, to the beginning of the first 5 minutes of persistent sleep.
Change from Baseline in the Mean Sleep Efficiency (SE) to Week 4 | From Baseline to Week 4 (28 days)
  Sleep Efficiency (SE) is measured as a range from 1 to 100. It is the percentage of the sleep period spent asleep (sleep total divided by sleep duration X 100%).
Change from Baseline in the Mean of Total Sleep Duration to Week 4 | From Baseline to Week 4 (28 days)
  Total sleep duration is measured objectively via an Oura ring. It is the total amount of sleep measured in seconds (total sleep duration = rem sleep +light sleep + deep sleep).
Change from Baseline in the Mean of Sleep Duration in Rapid Eye Movement (REM) to Week 4 | From Baseline to Week 4 (28 days)
  Sleep duration in REM is measured in seconds and objectively via an Oura ring. It is the total amount of REM sleep that is registered during the sleep period.
Change from Baseline in the Mean of Light Sleep Duration to Week 4 | From Baseline to Week 4 (28 days)
  Light Sleep Duration is measured in seconds and objectively via an Oura ring. It is the total amount of light sleep measured during the sleep period.
Change from Baseline in the Mean of Deep Sleep Duration to Week 4 | From Baseline to Week 4 (28 days)
  Deep sleep duration is measured in seconds and objectively via an Oura ring. It is the total amount of deep sleep registered during the sleep period.
Change from Baseline in the Mean Time in Bed to Week 4 | From Baseline to Week 4 (28 days)
  Time in bed is measured in seconds and objectively via an Oura ring. It is the total duration of the sleep period (Time in Bed = total sleep duration + awake time).
Change from Baseline in the Mean Heart Rate to Week 4 | From Baseline to Week 4 (28 days)
  Heart rate is the average heart rate registered during the sleep period via an Oura ring. It is measured in beats per minute.
Change from Baseline in the Mean Heart Rate Variability to Week 4 | From Baseline to Week 4 (28 days)
  Heart rate variability (HRV) is the average HRV calculated with RMSSD method via an Oura ring. It is measured in milliseconds.
Change from Baseline in the Mean of Respiratory Rate | From Baseline to Week 4 (28 days)
  Respiratory rate is measured objectively by an Oura ring. It is the average respiratory rate in breaths per minute.
Change from Baseline in the Mean Body Temperature to Week 4 | From Baseline to Week 4 (28 days)
  Body Temperature is measured objectively by an Oura ring. Body temperature, measured in Celsius, is the skin temperature deviation from the long-term temperature average.
Change from Baseline in the Mean of Daily Sleep Score to Week 4. | From Baseline to Week 4 (28 days)
  The Daily Sleep Score is composed of multiple sleep aspects collected by the Oura Ring, including deep sleep, rem sleep, efficiency, latency, restfulness, timing, and total sleep. Its score range is 0-100 (or Null if N/A).
  The Daily Sleep Score represents the overall sleep quality during the sleep period. It is calculated as a weighted average of sleep score contributors that each represent on aspect of sleep quality.
Change from Baseline in the Mean Daily Resilience Score to Week 4 | From Baseline to Week 4 (28 days)
  The Daily Resilience Score is composed of various data collected by the Oura ring, including sleep recovery, daytime recovery, and stress. The scores range from 1-100 (or Null if N/A).
Change from Baseline in the Mean of High Stress to Week 4 | From Baseline to Week 4 (28 days)
  High stress is the amount of stressed time in seconds that is calculated from stress samples detected by an Oura ring.
Change from Baseline in the Mean of High Recovery to Week 4 | From Baseline to Week 4 (28 days)
  High recovery is defined as the amount of recovery time in seconds calculated from stress samples identified by an Oura ring.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Goldenberg, ND, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No